CLINICAL TRIAL: NCT02426099
Title: Prevalence and Treatment of Resistant Hypertension in Diabetic Patients in Yaounde
Brief Title: Efficacy of Spironolactone in Cameroonian Diabetic Patients With Resistant Hypertension
Acronym: SPIRY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sobngwi Eugene (Other Government)
Collaborators: University of Yaounde 1 (Other)
Responsible Party: Sponsor-Investigator, Sobngwi Eugene, Professor and Consultant Physician, Yaounde Central Hospital
Organization: Yaounde Central Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNO22011
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension, Resistant to Conventional Therapy; Diabetes Mellitus
Keywords: Resistant hypertension; diabetes mellitus; Spironolactone; African
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Diabetes Mellitus | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose Spironolactone (Experimental): Add-on low dose 25 mg Spironolactone to current hypertension treatment
  Interventions: Drug: Low dose spironolactone
- Routine (Active Comparator): Routine intensification of anti hypertensive treatment based on existing guidelines
  Interventions: Other: Routine intensification of antihypertensive treatment

INTERVENTIONS:
Drug: Low dose spironolactone — 4-week add-on low dose spironolactone in resistant hypertension
  Other Names: Aldactone
  Arms: Low dose Spironolactone
Other: Routine intensification of antihypertensive treatment — 4-week guidelines oriented intensification of antihypertensive treatment
  Arms: Routine

SUMMARY:
This is a four-week randomized controlled single blinded trial of subjects presenting with resistant hypertension in a specialized diabetes care unit of Cameroon. They are randomly assigned using the method of blocks to treatment with a daily 25mg of spironolactone or to routine intensification of antihypertensive regimen , all added to previous regimen with unchanged diet. Visits are scheduled at the start of the treatment, at weeks two and four following add-on therapy initiation. The primary outcome is change in office and self-measurement blood pressure recorded at each visit, and secondary outcomes are variations in serum potassium, sodium, and creatinine levels.

ELIGIBILITY:
Inclusion Criteria:

* Resistant hypertension
* Diabetes mellitus

Exclusion Criteria:

* T2DM with overt acute/chronic complications,
* serum potassium ≥ 5.5 mmol/l,
* estimated Glomerular Filtration Rate (eGFR) calculated using the Modification of Diet in Renal Disease formula ≤ 30 ml/min/1.73m² of body weight,
* absolute contraindication to any of the drug regimen of the trial,
* and current aldosterone antagonist treatment or cessation within the last 15 months

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Efficacy (Blood pressure reduction) | 4 weeks
  Blood pressure reduction

SECONDARY OUTCOMES:
Potassium (Change in serum potassium) | 4 weeks
  Change in serum potassium
Creatinine (Change in serum creatinine) | 4 weeks
  Change in serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Mbanya, MD, PhD, Study Chair — University of Yaounde 1
Locations (1):
- National Obesity Centre, Yaounde Central Hospital, Yaoundé, Centre Region, Cameroon

REFERENCES:
- [Derived] Djoumessi RN, Noubiap JJ, Kaze FF, Essouma M, Menanga AP, Kengne AP, Mbanya JC, Sobngwi E. Effect of low-dose spironolactone on resistant hypertension in type 2 diabetes mellitus: a randomized controlled trial in a sub-Saharan African population. BMC Res Notes. 2016 Mar 23;9:187. doi: 10.1186/s13104-016-1987-5. PMID 27007793